CLINICAL TRIAL: NCT02623179
Title: Conventional and Molecular Diagnostic Method for Patients With Suspected Urinary Tract Infections: Clinical, Economic, and Quality of Life Outcomes
Brief Title: Conventional and Molecular Diagnostic Method for Patients With Suspected UTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Regional PCR, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PATUTI
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Urinary Tract Infections-UTI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-Culture and Sensitivity group (Active Comparator): Diagnosis by Culture and Sensitivity group-Treatment based on the results of the FH C & S testing - Odd Numbers on randomization table
  Interventions: Other: culture versus Molecular diagnostics
- B-Diagnosis by Molecular Testing (Active Comparator): Diagnosis by Molecular Testing-Treatment based on the results of the PathoGenius molecular testing - Even Numbers on randomization table
  Interventions: Other: culture versus Molecular diagnostics

INTERVENTIONS:
Other: culture versus Molecular diagnostics — Treatment based on the results of the FH C & S testing - Odd Numbers on randomization table

SUMMARY:
In this protocol, the investigators are examining the use of a novel pathogen testing technology and method of identification of antibiotic susceptibility against the conventional C & S testing for patients with both complicated and uncomplicated UTIs. The investigators will examine the two modes in terms of objective patient related outcomes, i.e. 1) diagnostic accuracy and degree of detail of final analysis; 2) time to resolution of symptoms; 3) quality of life as defined by particularly symptomology and "bothersomeness" of the symptoms; and 4) overall cost.

ELIGIBILITY:
Inclusion Criteria:

* • Age greater than or equal to 18 and less than or equal to 89 years.

  * The PI suspects the patient has a complicated or uncomplicated UTI that requires urine testing to confirm diagnosis
  * Able to provide at least 8 ml urine total (urine for 2 pathology tests).
  * Is willing to complete one follow up surveys and send back to FH.

Exclusion Criteria:

* • Unable or unwilling to provide written informed consent.

  * Unable to read and write English (surveys are not available or validated in any other language than English).
  * Currently on any antibiotic for any clinical indication.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
To quantify differences in the relative abundance and presence of microbial lineages as determined by culture and sequencing technologies. | 1 year
  comparison of culture and sensitivity results to the molecular results

SECONDARY OUTCOMES:
Time (as measured in hours) to preliminary and final identification of organism(s) and antibiotic sensitivity(s) results | 1 year
  time from collection of sample to diagnostic result delivery
Time from participant reported start of UTI symptoms to resolution. | 1 year
  collect time of reported UTI from Subject
Participant Quality of Life as measured by a UTI specific severity and bothersome of symptoms survey taken at baseline (at clinic visit) and at set time points post urine testing | 1 year
  collect data from Subject as outlined in the Quality of Life Assessment
Overall cost | 1 year
  collect data on the overall cost of Subject treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonald, MD, Principal Investigator — Florida Hospital Celebration Health